CLINICAL TRIAL: NCT00063622
Title: Clinical Research Network in Nonalcoholic Steatohepatitis: Pioglitazone vs. Vitamin E vs. Placebo for the Treatment of Non-Diabetic Patients With Nonalcoholic Steatohepatitis (PIVENS)
Brief Title: Pioglitazone vs Vitamin E vs Placebo for Treatment of Non-Diabetic Patients With Nonalcoholic Steatohepatitis (PIVENS)
Acronym: PIVENS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH - ADULT (IND); U01DK061730 (NIH)
Record Dates: First submitted 2003-07-01; First posted 2003-07-03 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2012-08

CONDITIONS: Liver Diseases
Keywords: Non alcoholic steatohepatitis; Steatohepatitis
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Pioglitazone; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Pioglitazone
  Interventions: Drug: Pioglitazone
- 2 (Active Comparator): Vitamin E
  Interventions: Dietary Supplement: Vitamin E
- 3 (Placebo Comparator): Placebo Pioglitazone or Placebo Vitamin E
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Pioglitazone — 30 mg daily
  Other Names: Actos
  Arms: 1
Dietary Supplement: Vitamin E — 800 IU daily
  Other Names: Nature Made
  Arms: 2
Drug: Matching placebo — Daily
  Arms: 3

SUMMARY:
The purpose of this study is to determine if therapy with pioglitazone or vitamin E will lead to an improvement in liver histology in non-diabetic adult patients with non-alcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
The purpose of this study is to determine if therapy with pioglitazone or vitamin E will lead to an improvement in liver histology in non-diabetic adult patients with non-alcoholic steatohepatitis (NASH).

ELIGIBILITY:
* Histologic evidence of NASH based on a liver biopsy obtained within 6 months of randomization.
* Age 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Shinde S, Nelson DR, Mitroi J, Heaton PC, Hincapie AL, Brouwers B. The roles of type 2 diabetes and obesity in disease activity and progression of non-alcoholic fatty liver disease/non-alcoholic steatohepatitis. Curr Med Res Opin. 2024 Jan;40(1):59-68. doi: 10.1080/03007995.2023.2279676. Epub 2024 Jan 3. PMID 37933187
- [Derived] Vilar-Gomez E, Gawrieh S, Liang T, McIntyre AD, Hegele RA, Chalasani N. Interrogation of selected genes influencing serum LDL-Cholesterol levels in patients with well characterized NAFLD. J Clin Lipidol. 2021 Mar-Apr;15(2):275-291. doi: 10.1016/j.jacl.2020.12.010. Epub 2020 Dec 27. PMID 33454241
- [Derived] Maev IV, Samsonov AA, Palgova LK, Pavlov CS, Shirokova EN, Vovk EI, Starostin KM. Effectiveness of phosphatidylcholine as adjunctive therapy in improving liver function tests in patients with non-alcoholic fatty liver disease and metabolic comorbidities: real-life observational study from Russia. BMJ Open Gastroenterol. 2020 Mar 26;7(1):e000368. doi: 10.1136/bmjgast-2019-000368. eCollection 2020. PMID 32337059
- [Derived] Kanwar P, Nelson JE, Yates K, Kleiner DE, Unalp-Arida A, Kowdley KV. Association between metabolic syndrome and liver histology among NAFLD patients without diabetes. BMJ Open Gastroenterol. 2016 Nov 9;3(1):e000114. doi: 10.1136/bmjgast-2016-000114. eCollection 2016. PMID 27933201
- [Derived] Corey KE, Vuppalanchi R, Wilson LA, Cummings OW, Chalasani N; NASH CRN. NASH resolution is associated with improvements in HDL and triglyceride levels but not improvement in LDL or non-HDL-C levels. Aliment Pharmacol Ther. 2015 Feb;41(3):301-9. doi: 10.1111/apt.13035. Epub 2014 Nov 28. PMID 25429853
- [Derived] Guy CD, Suzuki A, Abdelmalek MF, Burchette JL, Diehl AM; NASH CRN. Treatment response in the PIVENS trial is associated with decreased Hedgehog pathway activity. Hepatology. 2015 Jan;61(1):98-107. doi: 10.1002/hep.27235. Epub 2014 Aug 25. PMID 24849310
- [Derived] Hoofnagle JH, Van Natta ML, Kleiner DE, Clark JM, Kowdley KV, Loomba R, Neuschwander-Tetri BA, Sanyal AJ, Tonascia J; Non-alcoholic Steatohepatitis Clinical Research Network (NASH CRN). Vitamin E and changes in serum alanine aminotransferase levels in patients with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2013 Jul;38(2):134-43. doi: 10.1111/apt.12352. Epub 2013 May 29. PMID 23718573
- [Derived] Guerrerio AL, Colvin RM, Schwartz AK, Molleston JP, Murray KF, Diehl A, Mohan P, Schwimmer JB, Lavine JE, Torbenson MS, Scheimann AO. Choline intake in a large cohort of patients with nonalcoholic fatty liver disease. Am J Clin Nutr. 2012 Apr;95(4):892-900. doi: 10.3945/ajcn.111.020156. Epub 2012 Feb 15. PMID 22338037
- [Derived] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Derived] Chalasani NP, Sanyal AJ, Kowdley KV, Robuck PR, Hoofnagle J, Kleiner DE, Unalp A, Tonascia J; NASH CRN Research Group. Pioglitazone versus vitamin E versus placebo for the treatment of non-diabetic patients with non-alcoholic steatohepatitis: PIVENS trial design. Contemp Clin Trials. 2009 Jan;30(1):88-96. doi: 10.1016/j.cct.2008.09.003. Epub 2008 Sep 10. PMID 18804555
- See also: National Institute of Diabetes and Digestive and Kidney Diseases — http://www.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PIVENS enrollment started in January 2005 and ended in January 2007.
Pre-assignment Details: A total of 339 patients were registered and screened for PIVENS trial, 92 of whom (27%) were found ineligible. The failure to meet histological entry criteria and fasting blood glucose >125 mg/dL were the most frequent reasons for ineligibility.
Groups:
- Pioglitazone: Pioglitazone at a dose of 30 mg daily
- Vitamin E: Vitamin E at a dose of 800 IU daily
- Placebo: Placebo Pioglitazone and Placebo Vitamin E
Period: Overall Study
Arm/Group | Pioglitazone | Vitamin E | Placebo
Started | 80 | 84 | 83
Completed | 70 (All randomized patients were included in analysis of primary outcome) | 80 (All randomized patients were included in analysis of primary outcome) | 72 (All randomized patients were included in analysis of primary outcome)
Not Completed | 10 | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Vitamin E | Placebo | Total
Number analyzed (Participants) | 80 | 84 | 83 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.6) | 46.6 (12.1) | 45.4 (11.2) | 46.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 48 | 147
  Male | 33 | 32 | 35 | 100
Region of Enrollment [Number; unit: participants]
  United States | 80 | 84 | 83 | 247
Total nonalcoholic fatty liver disease (NAFLD) activity score [Mean (Standard Deviation); unit: scores on a scale] — Total nonalcoholic fatty liver disease (NAFLD) activity was assessed on a scale of 0 to 8, with higher scores indicating more severe disease; the components of this measure include steatosis (assessed on a scale of 0 to 3), lobular inflammation (assessed on a scale of 0 to 3), and hepatocellular ballooning (assessed on a scale of 0 to 2).
  scores on a scale | 5.0 (1.4) | 5.1 (1.4) | 4.8 (1.4) | 4.9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Non-alcoholic Fatty Liver Disease (NAFLD) Activity Defined by Change in Standardized Scoring of Liver Biopsies at Baseline and After 96 Weeks of Treatment.
Description: Total nonalcoholic fatty liver disease (NAFLD) activity was assessed on a scale of 0 to 8, with higher scores indicating more severe disease; the components of this measure include steatosis (assessed on a scale of 0 to 3), lobular inflammation (assessed on a scale of 0 to 3), and hepatocellular ballooning (assessed on a scale of 0 to 2). The primary outcome was an improvement in histological findings from baseline to 96 weeks, which required an improvement by 1 or more points in the hepatocellular ballooning score; no increase in the fibrosis score; and either a decrease in the activity score for nonalcoholic fatty liver disease to a score of 3 or less or a decrease in the activity score of at least 2 points, with at least a 1-point decrease in either the lobular inflammation or steatosis score.
Time Frame: baseline and 96 weeks
Population: All randomized participants were included in the analysis of the primary outcome.
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 80 | 84 | 83
participants | 27 | 36 | 16
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; The proportions in each active-treatment group (pioglitazone and vitamin E) in whom there was improvement in non-alcoholic steatohepatitis were compared with the proportion of subjects in the placebo group in whom there was improvement; Test type: Superiority or Other; p = 0.001, Mantel Haenszel — Given the fact that there were two planned primary comparisons, Bonferroni-adjusted P values of less than 0.025 were considered to indicate statistical significance
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.04, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Improvement in Steatosis
Description: Steatosis is assessed on a scale of 0 to 3 with higher scores indicating more severe steatosis. This secondary outcome measure is the number of participants that experienced a decrease in steatosis score, which indicates improvement in steatosis.
Time Frame: baseline and 96 weeks
Population: Number of subjects with biopsy specimens at baseline and 96 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 70 | 80 | 72
participants | 48 | 43 | 22
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.005, Fisher Exact
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Participants With Improvement in Lobular Inflammation
Description: Lobular inflammation is assessed on a scale of 0 to 3 with higher scores indicating more severe lobular inflammation. This secondary outcome measure is the number of participants that experienced a decrease in lobular inflammation score, which indicates improvement in lobular inflammation.
Time Frame: baseline and 96 weeks
Population: Number of subjects with biopsy specimens at baseline and 96 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 70 | 80 | 72
participants | 41 | 43 | 25
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.02, Fisher Exact
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.004, Fisher Exact

4. Secondary Outcome: Number of Participants With Improvement in Hepatocellular Ballooning
Description: Hepatocellular ballooning is assessed on a scale of 0 to 2 with higher scores indicating more severe hepatocellular ballooning. This secondary outcome measure is the number of participants that experienced a decrease in hepatocellular ballooning score, which indicates improvement in hepatocellular ballooning.
Time Frame: baseline and 96 weeks
Population: Number of subjects with biopsy specimens at baseline and 96 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 70 | 80 | 72
participants | 31 | 40 | 21
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.01, Fisher Exact
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.08, Fisher Exact

5. Secondary Outcome: Number of Participants With Improvement in Fibrosis
Description: Fibrosis is assessed on a scale of 0 to 4 with higher scores indicating more severe fibrosis. This secondary outcome measure is the number of participants that experienced a decrease in fibrosis score, which indicates improvement in fibrosis.
Time Frame: baseline and 96 weeks
Population: Number of subjects with biopsy specimens at baseline and 96 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 70 | 80 | 72
participants | 31 | 33 | 22
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.24, Fisher Exact
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.12, Fisher Exact

6. Secondary Outcome: Number of Participants With Resolution of Definite Nonalcoholic Steatohepatitis
Description: The criteria for nonalcoholic steatohepatitis was definite or possible steatohepatitis (assessed by a pathologist) with an activity score of 5 or more, or definite steatohepatitis (confirmed by two pathologists) with an activity score of 4. This secondary outcome measure is the number of participants who met this definition at baseline and did not meet this definition after 96 weeks of treatment and thus had a resolution of steatohepatitis.
Time Frame: baseline and 96 weeks
Population: Number of subjects with biopsy specimens at baseline and 96 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Vitamin E | Placebo
Number analyzed (Participants) | 70 | 80 | 72
participants | 33 | 29 | 15
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.001, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Vitamin E | Placebo
Serious Adverse Events (participants affected / at risk) | 2/80 | 7/84 | 10/83
Other Adverse Events (participants affected / at risk) | 41/80 | 46/84 | 40/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=80) | Vitamin E (N=84) | Placebo (N=83)
Severe adverse event (General disorders) | 2 | 7 | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=80) | Vitamin E (N=84) | Placebo (N=83)
Cardiovascular Event (Cardiac disorders) | 10 | 12 | 12
Bone fracture (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5
Diabetes (Endocrine disorders) | 0 | 4 | 0
Cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Other mild and moderate adverse event (General disorders) | 28 | 26 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No